CLINICAL TRIAL: NCT06067997
Title: Prevalence Of Pulmonary Embolism In Patients With HEmoptysis (POPEIHE)
Acronym: POPEIHE
Status: Completed | Type: Observational
Sponsor: Società Italiana di Medicina di Emergenza-Urgenza (Other)
Responsible Party: Sponsor
Other Study IDs: CEACV 20160118
Record Dates: First submitted 2023-09-12; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Hemoptysis; Pulmonary Embolism
MeSH Terms: conditions — Hemoptysis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pulmonary embolism diagnosis — The diagnosis of pulmonary embolism will be made using the diagnostic algorithm suggested by the 2019 European guidelines . The pre-test clinical probability of pulmonary embolism will be defined based on the simplified Wells score. In patients with a low pre-test clinical probability and a D-dimer level below the threshold value the diagnosis of pulmonary embolism will be excluded. The D-dimer level will be measured using the quantitative assay routinely used in each participating center; the threshold value for a positive result compared to a negative result is 500 μg per milliliter for patients under 50 years of age. For each additional decade of age, the exclusion cutoff will increase by 100 μg per milliliter.
  The criterion for the presence of pulmonary embolism is the detection of an intraluminal filling defect on CT.

SUMMARY:
Estimation of the incidence of pulmonary embolism in patients presenting to the Emergency Department with hemoptysis.

DETAILED DESCRIPTION:
Multicenter prospective observational cross-sectional study with non-commercial (non-profit) objectives.

The study population consists of consecutive patients who present to the Emergency Departments of the participating hospitals with hemoptysis.

The diagnosis of pulmonary embolism will be made using the diagnostic algorithm suggested by the 2019 European guidelines. The pre-test clinical probability of pulmonary embolism will be defined based on the simplified Wells score, which classifies pulmonary embolism as "likely" or "unlikely". In patients with a low pre-test clinical probability ("unlikely") and a D-dimer level below the threshold value (negative), the diagnosis of pulmonary embolism will be excluded, and further testing will not be necessary in this regard. The D-dimer level will be measured using the quantitative assay routinely used in each participating center; the threshold value for a positive result compared to a negative result is 500 μg per milliliter for patients under 50 years of age. For each additional decade of age, the exclusion cutoff will increase by 100 μg per milliliter.

For patients with a high pre-test clinical probability ("likely"), a positive D-dimer test, or both, a pulmonary CT angiography will be the diagnostic test of choice.

The criterion for the presence of pulmonary embolism is the detection of an intraluminal filling defect on CT.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who present to the Emergency Department of the participating centers with hemoptysis
* consent to participate.

Exclusion Criteria:

* Pregnancy.
* Age below 18 years.
* Terminal illnesses with an estimated prognosis of less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of consecutive patients who present to the Emergency Department of the participating hospitals with hemoptysis and agree to participate in the study. Patients under 18 years of age, pregnant patients, and patients with terminal illnesses with an estimated prognosis of less than 3 months will be excluded from the study. Data will be collected prospectively. The 30-day follow-up will be conducted by reviewing hospital documentation, any scheduled outpatient visits, any readmissions to the Emergency Department within the first 30 days in all Emergency Departments of the region, and, if necessary, through telephone follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
incidence of pulmonary embolism | 30 days within initial evaluation
  The incidence of pulmonary embolism in patients presenting to the Emergency Department with hemoptysis/haemoptysis.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Vanni, Professor, Study Chair — University of Florence
Locations (1):
- AOU Careggi, Florence, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hirshberg B, Biran I, Glazer M, Kramer MR. Hemoptysis: etiology, evaluation, and outcome in a tertiary referral hospital. Chest. 1997 Aug;112(2):440-4. doi: 10.1378/chest.112.2.440. PMID 9266882
- [Result] Vanni S, Bianchi S, Bigiarini S, Casula C, Brogi M, Orsi S, Acquafresca M, Corbetta L, Grifoni S. Management of patients presenting with haemoptysis to a Tertiary Care Italian Emergency Department: the Florence Haemoptysis Score (FLHASc). Intern Emerg Med. 2018 Apr;13(3):397-404. doi: 10.1007/s11739-017-1618-8. Epub 2017 Feb 3. PMID 28160237
- [Result] Larici AR, Franchi P, Occhipinti M, Contegiacomo A, del Ciello A, Calandriello L, Storto ML, Marano R, Bonomo L. Diagnosis and management of hemoptysis. Diagn Interv Radiol. 2014 Jul-Aug;20(4):299-309. doi: 10.5152/dir.2014.13426. PMID 24808437